CLINICAL TRIAL: NCT07062289
Title: Study on the Measurement of Portal Vein Pressure Gradient Guided by Endoscopic Ultrasound Based on Portal Vein Thrombosis and Portal Hypertension
Brief Title: Endoscopic Ultrasound-guided Measurement of Portal Vein Pressure Gradient
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaolong Zheng, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-0823
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Portal Vein Thrombosis; Portal Hypertension Related to Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hepatic venous pressure gradient, HVPG (Experimental): After puncturing the internal jugular vein, under the guidance of the image monitor, the balloon catheter is inserted into the hepatic vein along the blood vessel to measure the free hepatic venous pressure (FHVP), and then the balloon is inflated to measure the wedged hepatic venous pressure (WHVP). The difference between the two is the hepatic venous pressure gradient.
  Interventions: Procedure: endoscopic ultrasound-guided portal pressure gradient

INTERVENTIONS:
Procedure: endoscopic ultrasound-guided portal pressure gradient — This study employs an integrated endoscopic ultrasound-guided portal pressure gradient (EUS-PPG+) protocol uniquely designed for cirrhotic patients with portal vein thrombosis (PVT). Under general anesthesia in the left lateral decubitus position (novel positioning), a linear echoendoscope directs 22G needle puncture of the portal vein and inferior vena cava for direct pressure measurement, with real-time Doppler confirmation to avoid thrombosed vessels. Crucially, this intervention synchronizes diagnostic and therapeutic actions: if high-risk esophageal/gastric varices are identified during EUS, immediate endoscopic therapy (e.g., glue injection) is delivered in the same session. All participants additionally undergo standard hepatic venous pressure gradient (HVPG) measurement via transjugular access within 24 hours, enabling within-patient correlation analysis.

SUMMARY:
This study aims to evaluate the accuracy and safety of a novel endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) measurement technique in 42 adults with liver cirrhosis and portal vein thrombosis (blood clots in the liver's main vein), a condition where current standard testing (HVPG) fails to provide reliable pressure readings. Participants will undergo both EUS-PPG (using a specialized needle under ultrasound guidance) and HVPG procedures to compare results; EUS-PPG will be performed under general anesthesia in a left-side lying position-an innovative approach-while also enabling immediate endoscopic treatment of bleeding veins if detected during the same session. The primary goals are to validate EUS-PPG's safety in this high-risk group, establish its correlation with HVPG, and pioneer an integrated diagnosis-treatment protocol to reduce hospital stays and costs. The study runs from July 2025 to June 2027 at Zhejiang University School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* History of liver cirrhosis
* INR < 1.5
* Platelet count > 50 × 10⁹/L
* Patients agreed to HVPG and EUS-PPG measurements

Exclusion Criteria:

* Patients with ascites
* Patients with renal insufficiency
* Patients with active infection
* Patients with hepatic encephalopathy
* Critically ill patients
* Pregnant patients
* Patients with immunodeficiency diseases (such as systemic lupus erythematosus)
* Patients with mental illness
* Patients with malignant tumors
* Patients who refused to undergo HVPG and EUS-PPG measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Portal Pressure Gradient Measured by HVPG and EUS-PPG Techniques | From enrollment, treatment was completed within 1 week
  The internal jugular vein is punctured and the difference between the wedge hepatic venous pressure (WHVP) and the free hepatic venous pressure (FHVP) is measured as the hepatic venous pressure gradient (HVPG). Endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) refers to the measurement of data by passing the puncture needle through the digestive tract into the portal vein system, hepatic vein or inferior vena cava system under the guidance of a linear array ultrasound endoscope.Portal vein pressure (PVP): The normal portal vein pressure is 1.27-2.35 kPa (13-24 cmH2O)

SECONDARY OUTCOMES:
Incidence of surgery-related complications | From enrollment, treatment was completed within 1 week
  Complications: obvious abdominal pain and nausea, fever > 38.5°C
Direct medical cost of treatment | From enrollment, treatment was completed within 1 week
  Direct medical cost of treatment:
  Components: surgical consumables, anesthesia, drugs, ward fees, nursing Currency: RMB (yuan)

IPD SHARING:
Plan to Share IPD: No
The patient's basic data and information will be kept confidential

REFERENCES:
- [Result] Martinez-Moreno B, Martinez Martinez J, Herrera I, Guilabert L, Rodriguez-Soler M, Bellot P, Miralles C, Pascual S, Irurzun J, Zapater P, Palazon-Azorin JM, Gil Guillen V, Jover R, Aparicio JR. Correlation of endoscopic ultrasound-guided portal pressure gradient measurements with hepatic venous pressure gradient: a prospective study. Endoscopy. 2025 Jan;57(1):62-67. doi: 10.1055/a-2369-0759. Epub 2024 Jul 18. PMID 39025130
- [Result] Zhang W, Peng C, Zhang S, Huang S, Shen S, Xu G, Zhang F, Xiao J, Zhang M, Zhuge Y, Wang L, Zou X, Lv Y. EUS-guided portal pressure gradient measurement in patients with acute or subacute portal hypertension. Gastrointest Endosc. 2021 Mar;93(3):565-572. doi: 10.1016/j.gie.2020.06.065. Epub 2020 Jun 29. PMID 32615178